CLINICAL TRIAL: NCT01479348
Title: Phase 0 Trial of [F-18]-5-Fluoro-2'-Deoxycytidine With Tetrahydrouridine
Brief Title: Imaging Study for FdCyd and THU Cancer Treatment
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow, insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Choyke, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 120014; 12-C-0014
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms
Keywords: Imaging; Radiopharmaceutical; Safety; Dosimetry; Drug Distribution; Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Neoplasms | interventions — Tetrahydrouridine; Positron-Emission Tomography; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1/Intravenous (IV) Tetrahydrouridine (THU) (Experimental): [F-18]-5-fluoro-2'-deoxycytidine plus Tetrahydrouridine
  Interventions: Drug: [F-18]-5-FLUORO-2'-DEOXYCYTIDINE; Drug: Tetrahydrouridine intravenous (IV); Drug: Tetrahydrouridine (oral); Diagnostic Test: Positron emission tomography (PET)/Computed tomography (CT)
- 2/Oral Tetrahydrouridine (THU) (Experimental): [F-18]-5-fluoro-2'-deoxycytidine plus Tetrahydrouridine
  Interventions: Drug: [F-18]-5-FLUORO-2'-DEOXYCYTIDINE; Drug: Tetrahydrouridine intravenous (IV); Drug: Tetrahydrouridine (oral); Diagnostic Test: Positron emission tomography (PET)/Computed tomography (CT)

INTERVENTIONS:
Drug: [F-18]-5-FLUORO-2'-DEOXYCYTIDINE — 18FdCyd radiotracer
  Other Names: 18FdCyd
Drug: Tetrahydrouridine intravenous (IV) — Total dose of THU = 350 mg/m^2, IV
  Other Names: THU
Drug: Tetrahydrouridine (oral) — Total dose of THU is 3000 mg, oral
  Other Names: THU
Diagnostic Test: Positron emission tomography (PET)/Computed tomography (CT) — One prior CT and 3 sequential whole body PET
  Other Names: PET scan/CT scan

SUMMARY:
Background:

- The drugs FdCyd (also called 5-fluoro-2'-deoxycytidine) and THU (also called tetrahydrouridine) are being used in a cancer treatment study. Not a lot is known about how FdCyd works in the body. Researchers want to look at a modified form of FdCyd using imaging studies to see how the drug reacts with the cancer. This study is not a treatment study. It is open only to people who are already on the FdCyd and THU cancer treatment study.

Objectives:

- To study how FdCyd affects advanced cancer cells.

Eligibility:

- Participants in National Cancer Institute study 09-C-0214.

Design:

* Participants will have two imaging studies, one before starting FdCyd and THU treatment and one after starting treatment.
* Participants will have the modified FdCyd, known as F-18 FdCyd, with a dose of THU. The doses will be followed by two imaging study scans and frequent blood samples.
* This procedure will be repeated at a later date, during the FdCyd and THU treatment period.
* Treatment will not be provided as part of this study. This is an imaging study protocol only....

DETAILED DESCRIPTION:
BACKGROUND:

- In pre-clinical models, 5-fluoro-2-deoxycytidine (FdCyd), administered along with

tetrahydrouridine (THU; an inhibitor of cytidine/deoxycytidine deaminase), has shown superior anti-tumor activity as compared with 5-fluorouracil.

- FdCyd can be phosphorylated to 5-fluoro-2-deoxycytidylate (FdCMP) by deoxycytidine

kinase and the nucleotide deaminated to FdUMP by deoxycytidylate (dCMP) deaminase.

The activity of dCMP deaminase is reported to be higher in human malignancies than in normal tissues, which may result in selective cytotoxicity.

* FdCyd is an inhibitor of deoxyribonucleic acid (DNA) methyltransferase and DNA methylation, resulting in reexpression of genes silenced by DNA hypermethylation. It is being evaluated in a phase II multihistology clinical trial at the Developmental Therapeutics Clinic, National Cancer Institute (NCI), Clinical Center, National Institutes of Health (NIH).
* While FdCyd + THU has shown preliminary evidence of activity in early phase trials not all patients show clinical response. The establishment of a radiolabeled form to image the biodistribution in vivo at baseline and during therapy may provide insight into the distribution of the therapeutic drug.
* The first step in the development of such an in vivo marker is to determine the

biodistribution and safety of the radiolabeled form.

OBJECTIVES:

* Determine the safety of [F-18]-5-fluoro-2'-deoxycytidine (FdCyd) administered intravenously with administration of tetrahydrouridine (THU).
* Estimate the radiation dosimetry of [F-18]-FdCyd in humans.

ELIGIBILITY:

* Only patients enrolled in NCI Phase II Study evaluating FdCyd with THU (NCI Protocol # 09-C-0214 (CTEP# 8351) or NCI Protocol #12-C-0066 (CTEP# 9127)) at the NIH Clinical Center will be eligible to participate in this study).
* Patients must have a target lesion greater than or equal to 10mm
* May not be pregnant or lactating; must be less than or equal to 350 lbs; and may not have known allergy to FdCyd or contraindications to positron emission tomography (PET)/computed tomography (CT) imaging.

DESIGN:

* There are two arms to this study
* The first arm will be patients enrolling in the therapeutic Phase II 5-FdCyd/THU study (NCI Protocol # 09-C-0214 (CTEP# 8351) in the NCI Developmental Therapeutics Clinic
* The second arm will be patients enrolling in the Phase I 5-FdCyd/THU study (NCI Protocol #12-C-0066 (CTEP# 9127)) in the NCI Developmental Therapeutics Clinic.
* Patients will undergo an initial [F-18]-FdCyd + THU PET/CT imaging prior to therapeutic dosing on study NCI Protocol # 09-C-0214 (CTEP# 8351) or NCI Protocol #12-C-0066 (CTEP# 9127). Repeat imaging will be performed while the patient is receiving FdCyd + THU therapy under the parent therapeutic protocol. This imaging must be completed 2-5 days after cycle start and at least 2 hours after a dose. Upon completion of repeat imaging, patients will be taken off this imaging study 24 hours after the last imaging session.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Enrolled in the National Institutes of Health (NIH) Phase II Clinical protocol evaluating 5-fluro-2'-deoxycytidine (FdCyd) with Tetrahydrouridine (THU) (09-C-0214) with target lesion measured as greater than or equal to 10mm with spiral computed tomography (CT) scan.
* Written, voluntary, informed consent of the patient must be obtained in compliance with institutional, state and federal guidelines
* For females: Negative serum pregnancy test OR post-menopausal for at least 2 years OR patient has had a hysterectomy

EXCLUSION CRITERIA:

* Participants with severe claustrophobia unresponsive to oral anxiolytics
* Subjects weighing > 400 lbs (weight limit for scanner table), or unable to fit within the imaging gantry
* Known allergy to FdCyd
* The subject is unable to lie still for 75 minutes
* 5 Pregnant or lactating women. Pregnant women are excluded from this study because the effects of 18F-FdCyd in pregnancy are not known. Because there is an unknown but potential risk for adverse events in nursing infants secondary to administration of 18F-FdCyd in the mother, breastfeeding should be discontinued if the mother receives 18F-FdCyd
* Participants with any co-existing medical or psychiatric condition that is likely to interfere with study procedures and/or results

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Kurdziel, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carter SK. Editorial: Large-bowel cancer-The current status of treatment. J Natl Cancer Inst. 1976 Jan;56(1):3-10. doi: 10.1093/jnci/56.1.3. No abstract available. PMID 1255749
- [Background] Doroshow JH, Multhauf P, Leong L, Margolin K, Litchfield T, Akman S, Carr B, Bertrand M, Goldberg D, Blayney D, et al. Prospective randomized comparison of fluorouracil versus fluorouracil and high-dose continuous infusion leucovorin calcium for the treatment of advanced measurable colorectal cancer in patients previously unexposed to chemotherapy. J Clin Oncol. 1990 Mar;8(3):491-501. doi: 10.1200/JCO.1990.8.3.491. PMID 2407810
- [Background] HARTMANN JR, ORIGENES ML Jr, MURPHY ML, SITARZ A, ERLANDSON M. EFFECTS OF 2'-DEOXY-5-FLUOROURIDINE (NSC-27640) AND 5-FLUOROURACIL (NSC-19893) ON CHILDHOOD LEUKEMIA. Cancer Chemother Rep. 1964 Jan;34:51-4. No abstract available. PMID 14116219

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled in the 2/Oral Tetrahydrouridine (THU) Group.
Period: Overall Study
Arm/Group | 1/Intravenous (IV) Tetrahydrouridine (THU) | 2/Oral Tetrahydrouridine (THU)
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1/Intravenous (IV) Tetrahydrouridine (THU): [F-18]-5-fluoro-2'-deoxycytidine plus Tetrahydrouridine
  [F-18]-5-FLUORO-2'-DEOXYCYTIDINE: 18FdCyd radiotracer
  Tetrahydrouridine intravenous (IV): Total dose of Tetrahydrouridine (THU) = 350 mg/m^2, IV
  Tetrahydrouridine (oral): Total dose of THU is 3000 mg, oral
  Positron emission tomography (PET)/Computed tomography (CT): One prior CT and 3 sequential whole body PET
Arm/Group | 1/Intravenous (IV) Tetrahydrouridine (THU)
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.46 (15.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Baseline Tumor Types [Count of Participants; unit: Participants]
  Head & Neck Carcinoma | 2
  Non-Small Cell Lung Carcinoma | 2
  Hepatocellular Carcinoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Description: [F-18]-5-fluoro-2'-deoxycytidine (FdCyd) was administered intravenously with administration of tetrahydrouridine (THU) and the frequency and severity of adverse events was observed. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 0 is normal, Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe or medically significant but not immediately life-threatening, Grade 4 is life-threatening consequences, and Grade 5 is death related to adverse event.
Time Frame: Within 5 days after interventions
Measure: Number; unit: adverse events
Arm/Group | 1/Intravenous (IV) Tetrahydrouridine (THU)
Number analyzed (Participants) | 5
adverse events
  Day 1 Adverse Events | 0
  Day 2, Grade 2 Hypoalbuminemia | 1
  Day 2, Grade 3 Anemia | 1
  Day 3 Adverse Events | 0
  Day 4 Adverse Events | 0
  Day 5 Adverse Events | 0

2. Primary Outcome: Radiation Dosimetry Estimates of 5-fluoro-2'-Deoxycytidine (FdCyd) in Humans
Description: Radiation dosimetry was determined based on the first patients. This involved making region of interest measurements on the scan for each major organ and measuring the uptake. Using standard dosimetry software this is converted into mSv/MBq, a standard measure of dosimetry. The software is known as Organ Level INternal Dose Assessment/EXponential Modeling (OLINDA) and is commonly used to generate this kind of data.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | 1/Intravenous (IV) Tetrahydrouridine (THU)
Number analyzed (Participants) | 5
mSv/MBq
  Adrenals | 1.83 (9.3)
  Brain | 8.17 (2.04)
  Breasts | 1.03 (1.01)
  Gallbladder wall | 4.05 (7.55)
  Lower large intestine wall | 2.52 (7.82)
  Small intestine | 2.13 (4.57)
  Stomach wall | 1.90 (3.27)
  Upper large intestine wall | 2.04 (6.43)
  Heart wall | 1.10 (1.82)
  Kidneys | 5.26 (2.23)
  Liver | 6.02 (2.74)
  Lungs | 1.82 (7.10)
  Muscle | 1.16 (1.35)
  Ovaries | 1.57 (2.22)
  Pancreas | 1.63 (4.27)
  Red marrow | 1.14 (2.19)
  Osteogenic cells | 1.71 (6.41)
  Skin | 8.65 (1.19)
  Spleen | 1.69 (5.55)
  Testes | 1.03 (2.38)
  Thymus | 1.12 (3.01)
  Thyroid | 8.23 (4.39)
  Urinary bladder wall | 7.96 (5.24)
  Uterus | 1.63 (4.99)

3. Secondary Outcome: Tumor to Background Ratios (TBRs) of Target Lesions at 4 Time Points After Injection
Description: Participants were scanned by positron emission tomography (PET) and lesions were measured at 4 time points after injection.
Time Frame: 9 minutes, 32 minutes, 56 minutes and 2 hours after injection
Population: One participant contributed to data in each row.
Measure: Number; unit: TBR ratio
Arm/Group | 1/Intravenous (IV) Tetrahydrouridine (THU)
Number analyzed (Participants) | 5
TBR ratio
  Pt 1 L. Parotid adenosquam. cell ca at 9 min: number analyzed (Participants) | 1
  Pt 1 L. Parotid adenosquam. cell ca at 9 min | 1.4
  Pt 1 L. Parotid adenosquam. cell ca at 32 min: number analyzed (Participants) | 1
  Pt 1 L. Parotid adenosquam. cell ca at 32 min | 1.5
  Pt 1 L. Parotid adenosquam. cell ca at 56 min: number analyzed (Participants) | 1
  Pt 1 L. Parotid adenosquam. cell ca at 56 min | 1.5
  Pt 1 L. Parotid adenosquam. cell ca at 2 hrs: number analyzed (Participants) | 1
  Pt 1 L. Parotid adenosquam. cell ca at 2 hrs | 1.6
  Pt 2 R. Parapharyngeal Spindle Cell Ca at 9 min: number analyzed (Participants) | 1
  Pt 2 R. Parapharyngeal Spindle Cell Ca at 9 min | 1.9
  Pt 2 R. Parapharyngeal Spindle Cell Ca at 32 min: number analyzed (Participants) | 1
  Pt 2 R. Parapharyngeal Spindle Cell Ca at 32 min | 1.7
  Pt 2 R. Parapharyngeal Spindle Cell Ca at 56 min: number analyzed (Participants) | 1
  Pt 2 R. Parapharyngeal Spindle Cell Ca at 56 min | 1.7
  Pt 2 R. Parapharyngeal Spindle Cell Ca at 2 hrs: number analyzed (Participants) | 1
  Pt 2 R. Parapharyngeal Spindle Cell Ca at 2 hrs | 1.6
  Pt 3 Non-small Cell Lung Ca at 9 min: number analyzed (Participants) | 1
  Pt 3 Non-small Cell Lung Ca at 9 min | 1.4
  Pt 3 Non-small Cell Lung Ca at 32 min: number analyzed (Participants) | 1
  Pt 3 Non-small Cell Lung Ca at 32 min | 1.4
  Pt 3 Non-small Cell Lung Ca at 56 min: number analyzed (Participants) | 1
  Pt 3 Non-small Cell Lung Ca at 56 min | 1.5
  Pt 3 Non-small Cell Lung Ca at 2 hrs: number analyzed (Participants) | 1
  Pt 3 Non-small Cell Lung Ca at 2 hrs | 1.7
  Pt 4 Non-small Cell Lung Ca at 9 min: number analyzed (Participants) | 1
  Pt 4 Non-small Cell Lung Ca at 9 min | 2.4
  Pt 4 Non-small Cell Lung Ca at 32 min: number analyzed (Participants) | 1
  Pt 4 Non-small Cell Lung Ca at 32 min | 2.1
  Pt 4 Non-small Cell Lung Ca at 56 min: number analyzed (Participants) | 1
  Pt 4 Non-small Cell Lung Ca at 56 min | 1.6
  Pt 4 Non-small Cell Lung Ca at 2 hrs: number analyzed (Participants) | 1
  Pt 4 Non-small Cell Lung Ca at 2 hrs | 2.0
  Pt 5 Hepatocellular Ca at 9 min: number analyzed (Participants) | 1
  Pt 5 Hepatocellular Ca at 9 min | NA — Activity within the tumor was not clearly discernable from remainder of liver parenchyma, thus TBRs are not included for Pt. 5 because of concern about reporting misleading values in setting of high background/surrounding liver uptake.
  Pt 5 Hepatocellular Ca at 32 min: number analyzed (Participants) | 1
  Pt 5 Hepatocellular Ca at 32 min | NA — Activity within the tumor was not clearly discernable from remainder of liver parenchyma, thus TBRs are not included for Pt. 5 because of concern about reporting misleading values in setting of high background/surrounding liver uptake.
  Pt 5 Hepatocellular Ca at 56 min: number analyzed (Participants) | 1
  Pt 5 Hepatocellular Ca at 56 min | NA — Activity within the tumor was not clearly discernable from remainder of liver parenchyma, thus TBRs are not included for Pt. 5 because of concern about reporting misleading values in setting of high background/surrounding liver uptake.
  Pt 5 Hepatocellular Ca at 2 hrs: number analyzed (Participants) | 1
  Pt 5 Hepatocellular Ca at 2 hrs | NA — Activity within the tumor was not clearly discernable from remainder of liver parenchyma, thus TBRs are not included for Pt. 5 because of concern about reporting misleading values in setting of high background/surrounding liver uptake.

4. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 20 months and 12 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Intravenous (IV) Tetrahydrouridine (THU)
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 20 months and 12 days.
Arm/Group | 1/Intravenous (IV) Tetrahydrouridine (THU)
All-Cause Mortality (participants affected / at risk) | 2/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Intravenous (IV) Tetrahydrouridine (THU) (N=5)
Death NOS (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Intravenous (IV) Tetrahydrouridine (THU) (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2015-03-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT01479348/Prot_SAP_000.pdf
  • Informed Consent Form: IV FdCyd + THU (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT01479348/ICF_001.pdf
  • Informed Consent Form: Oral FdCyd + THU (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/48/NCT01479348/ICF_002.pdf